CLINICAL TRIAL: NCT06750549
Title: Mobile Application for Patient Engagement and Physician-Directed Remote Management of Heart Failure: The ENGAGE-HF Study
Brief Title: Mobile Application for Patient Engagement and Physician-Directed Remote Management of Heart Failure
Acronym: ENGAGE-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Stanford University (Other); Johns Hopkins University (Other); Boston University (Other)
Responsible Party: Principal Investigator, Michael Dorsch, Associate Professor of Pharmacy, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00240067
Record Dates: First submitted 2024-12-11; First posted 2024-12-27 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
Keywords: Medication Optimization
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: 1:1 randomization by site
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The ENGAGE-HF intervention is a combination of a patient-facing mobile application that is integrated with a remote blood pressure cuff and scale along with a clinician-facing dashboard. The mobile application helps complete standard ambulatory monitoring recommended by heart failure clinicians. Simultaneously, the application includes visualizations of that data and education for patients that is intended to promote patient engagement and patient understanding of heart failure care. The information is then made available to treating clinicians via a PDF summary to facilitate outpatient management of the patient by the clinician. There are also a select set of notifications triggered by the ENGAGE-HF platform that will be transmitted to the treating clinician.
  Interventions: Device: ENGAGE-HF Mobile Application
- Control Group (No Intervention): Participants randomized to the control group will receive usual heart failure care.

INTERVENTIONS:
Device: ENGAGE-HF Mobile Application — The mobile app aids ambulatory heart failure monitoring and patient engagement through several features:
  Physiologic Monitoring: Daily tracking of blood pressure, weight, and heart rate using Bluetooth devices. Data is shown in graphical and tabular formats.
  Health Status Assessment: Biweekly KCCQ-12 surveys and dizziness questions provide scores (0-100), helping visualize therapy benefits and medication adherence, and reducing clinician inertia.
  Medication Checklist: Lists current medications and target doses for common heart failure therapies, encouraging adherence and optimization, with alerts for potential improvements.
  Education: Animated videos from heart failure experts and societies explain medications, monitoring rationale, app features, and interpretation of data.
  The app enhances heart failure management via consistent monitoring, assessment, medication adherence, and educational content.
  Arms: Intervention

SUMMARY:
The ENGAGE-HF mobile application tracks three key features over time: (1) heart failure health status, (2) vital signs (e.g., blood pressure, heart rate) and weight, and (3) the quality of heart failure medication therapy. Helping patients understand how these characteristics interact and change over time may improve their ability to understand and manage heart failure.

In this study, the investigators aim to evaluate whether the ENGAGE-HF mobile application, by facilitating the behavior change strategies of self-monitoring and feedback, and a clinician-facing dashboard, improves the optimization of heart failure guideline-directed medical therapies (GDMT) and quality of life.

An optional sub-study of cognitive function will invite all eligible participants enrolled in the main study to participate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure
* Last left ventricular ejection fraction within 2 years < 50% based on echocardiogram, MRI, CT, or nuclear perfusion and, if no ejection fraction documented, then clinical documentation of heart failure with reduced ejection fraction
* Currently admitted with upcoming discharge or discharged from hospital within the prior 4 weeks
* At least two eligible heart failure therapies (guideline-recommended BB, RASI, MRA, or SGLT2i) not yet initiated or at < 50% of target dose at time of enrollment

Exclusion Criteria:

* Receives dialysis
* Inotropic therapy after hospitalization
* History of a prior solid organ transplant or actively listed on heart transplant waiting list
* History of left ventricular assist device implantation
* Cardiac amyloidosis
* Currently pregnant or intends to become pregnant during the study period
* Life expectancy estimated less than 6 months related to cardiac or non-cardiac comorbidities as per investigator's judgment
* Actively enrolled in hospice or comfort care
* Currently participating in an investigational device or drug study or having participated in such a study 30 days prior to screening
* Subject without a compatible smartphone
* Subject not proficient with written and spoken English
* Any other disorder or condition that, in the opinion of the investigator would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Participant has diminished decision-making capacity
* Admitted to or planned discharge to a skilled nursing facility or rehabilitation facility (acute or subacute)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Medication optimization score at 90 days | From enrollment to the end of participation at 90 days
  The primary outcome will be the difference in the medication optimization score at 90 days between the intervention and control group. The MOS is a percent between 0 (least optimized) and 100 (most optimized), which represents the extent of medication optimization that needs to be performed. Inputs for the score include medications, vital signs, and laboratory values, and thus, the score accounts for contraindications to medical therapy titration. The score has been shown to correlate with clinical outcomes in two large randomized controlled trials.

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ-23) | Baseline and at 90 days
  The secondary outcome will be heart failure symptoms as assessed by the difference between the intervention and the control groups in the 23-item Kansas City Cardiomyopathy Questionnaires (KCCQ-23) clinical summary score at 90 days.
  The KCCQ-23 quantifies patients' health status over the prior 2 weeks and has extensive data supporting its validity, reliability, and sensitivity to clinical change. Scores will be transformed into a 0-100 point rating, with lower scores representing worse health status.

OTHER OUTCOMES:
Kansas City Medical Optimization (KCMO) score | From enrollment to the end of participation at 90 days
  Kansas City Medical Optimization (KCMO) is the average total daily dose for each eligible Guideline-Directed Medical Therapy (GDMT) drug class divided by its target dose. The investigators will compare this score with the primary outcome measure.
Modified Continuous 4-Pillar Score | From enrollment to the end of participation at 90 days
  The Modified Continuous 4-Pillar Score (C4P) score is a continuous version of the 4P Intensification Score, where each dose escalation leads to an increase in the score rather than assigning the same points to a range of increasing GDMT doses. For Beta Blockers, ACEI/ARBs, MRAs, and SGLT2 inhibitor, the C4P score is calculated as 2 + 2 × (% of target daily dose) for patients on therapy to a max score of 4. For ARNI therapy, the score is calculated as 4 + 2 × (% of target daily dose). The score range is from 0 to 18. A higher score is a better outcome.
90 day all-cause mortality | From enrollment to the end of participation at 90 days
  Participant deaths
Heart failure hospitalization | From enrollment to the end of participation at 90 days
  Participant hospitalization due to heart failure. Heart failure hospitalizations will be defined as outlined by the Heart Failure Collaboratory and Academic Research Consortium
Emergency department visits for heart failure | From enrollment to the end of participation at 90 days
  Participant visits to the emergency department for heart failure. Emergency department visits will use a modified version of the criteria of the Heart Failure Collaboratory and Academic Research Consortium without the 24 hour hospital admission requirement.
Outpatient intravenous diuresis | From enrollment to the end of participation at 90 days
  Participant undergoes outpatient intravenous diuresis.
Process measures | From enrollment to the end of participation at 90 days
  The investigators will evaluate process measures related to use of the intervention and downstream clinical processes. This will include patient engagement with the ENGAGE-HF mobile application and the subcomponents of engagement with respect to the different aspects of the mobile application.
Mini-Cog Cognitive Assessment | At baseline
  The Mini-Cog is a brief screening tool used to assess cognitive function, particularly memory and executive function, in study participants. The assessment consists of two components: a three-item recall test and a clock-drawing test (CDT). The three-item recall test evaluates short-term memory by requiring participants to remember and later recall three unrelated words. The CDT assesses executive function and visual-spatial skills by requiring participants to draw a clock with a specified time.
Memory Recall - Immediate | Baseline and at 90 days
  In the Memory Recall - Immediate part of the INTACT neurocognitive assessment, participants recall and select five animal names. Measured by the average number of correct responses (0-5) and completion time (seconds).
Choice Reaction Time | Baseline and at 90 days
  In the Choice Reaction Time part of the INTACT neurocognitive assessment, participants identify the direction of an arrow in an odd-colored block among three. Measured by the proportion of correct responses (true/false) and average reaction time (seconds).
Visual Paired Associates | Baseline and at 90 days
  In the Visual Paired Associates part of the INTACT neurocognitive assessment, participants match image pairs after learning them. Measured by the proportion of correct responses (true/false) and average reaction time (seconds).
Digit Symbol Matching | Baseline and at 90 days
  In the Digit Symbol Matching part of the INTACT neurocognitive assessment, participants match symbols to numbers using a reference. Measured by the proportion of correct responses (true/false) and average reaction time (seconds).
Spatial Memory | Baseline and at 90 days
  In the Spatial Memory part of the INTACT neurocognitive assessment, participants recreate increasingly complex block designs. Measured by the proportion of correct responses (true/false) and average reaction time (seconds).
Memory Recall - Delayed | Baseline and at 90 days
  In the Memory Recall - Delayed part of the INTACT neurocognitive assessment, participants recall the five animal names from the immediate recall test after a delay. Measured by the average number of correct responses (0-5) and completion time (seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dorsch, PharmD, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - Stanford Cardiovascular Clinic, Stanford, California
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - U-M Frankel Cardiovascular Center, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Undecided